CLINICAL TRIAL: NCT03744533
Title: Head-down Position for Acute Ischemic Stroke With Large Artery Atherosclerosis: a Prospective, Random, Multi-Center, Pilot Trial
Brief Title: Head-down Position for Acute Ischemic Stroke With Large Artery Atherosclerosis
Acronym: HOPES2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Department Chairman, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: k （2018）38
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Ischemic Stroke
Keywords: head-down position; Large Artery Atherosclerosis
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- head-down position treatment (Experimental)
  Interventions: Other: head-down position treatment; Other: guideline-based treatment
- guideline-based treatment (Active Comparator)
  Interventions: Other: guideline-based treatment

INTERVENTIONS:
Other: head-down position treatment — the head position of subjects is lowered to 20 degrees in a supine position between 8:00-22:00 within 24h post-randomization as long as possible. During the procedure, when subjects feel intolerable, the head position will be elevated to lying flat (0 degree) for 5-10min, and then the above procedure is repeated. After 24h post-randomization, the head down procedures with -20 degrees in a supine position with duration of 1-1.5 hour will be performed three times daily at 9:00-11:00, 15:00-17:00 and 20:00-22:00, respectively.
  Arms: head-down position treatment
Other: guideline-based treatment — guideline-based treatment

SUMMARY:
Currently, the guideline recommended re-perfusion such as intravenous thrombolysis and mechanical thrombectomy as the most effective treatment for acute ischemic stroke. However, the two methods are restricted by a strict time window, which greatly limits the number of the patients receiving treatment. The abundant studies have suggested that good collateral circulation can provide compensatory blood supply to save the ischemic penumbra and reduces the infarct volume, which improves the prognosis. How to improve collateral circulation in an efficient and safe way is a clinical challenge. Our recent experiment results of the animal and preliminary clinical experiments show that head-down position may significantly increase cerebral perfusion and improve neurological function. Clinically, head-down position is simple and easy to operate, and theoretically may increases brain perfusion and improve collateral circulation. A pilot randomized clinical trial is designed to investigate the effect of head-down position combined with routine rehabilitation in patients with ischemic stroke.The study is designed to explore the efficacy and safety of head-down position in patients with acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Patient age over 18 years
2. acute ischemic stroke within 24 h of onset
3. neurological deficit: 6≤NIHSS≤16
4. Large artery atherosclerosis etiology based on TOAST typing
5. the supplied vessel is the middle cerebral artery or internal carotid artery, and the degree of stenosis was more than 50%.
6. first stroke onset or past stroke without obvious neurological deficit (mRS≤1)
7. Signed informed consent

Exclusion Criteria:

1. Disturbance of consciousness
2. Hemorrhagic stroke or mixed stroke
3. Combining with severe organ dysfunction
4. Past hemorrhagic stroke
5. A history of stroke with severe sequelae
6. Planned revascularization within 3 months
7. Ischemic stroke due to surgical intervention
8. participating in other clinical trials within 3 months
9. Pregnant or lactating women
10. any inappropriate patient assessed by the researcher

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2021-08-28 (Actual); Study Completion 2021-08-28 (Actual)

PRIMARY OUTCOMES:
proportion of modified Rankin Score of 0 to 2 | 90 days

SECONDARY OUTCOMES:
Proportion of modified Rankin Score of 0 to 1 | 90 days
proportion of early neurological deterioration | 48 hours
  Early neurological deterioration, defined as more than 4 increase in National Institute of Health stroke scale score
The occurence of stroke or other vascular events | 90 days
proportion of death of any cause | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Huisheng Chen, Doctor, Study Chair — Neurology Department
Locations (1):
- General Hospital of ShenYang Military Region, Shenyang, China

REFERENCES:
- [Derived] Chen HS, Zhang NN, Cui Y, Li XQ, Zhou CS, Ma YT, Zhang H, Jiang CH, Li RH, Wan LS, Jiao Z, Xiao HB, Li Z, Yan TG, Wang DL, Nguyen TN. A randomized trial of Trendelenburg position for acute moderate ischemic stroke. Nat Commun. 2023 May 5;14(1):2592. doi: 10.1038/s41467-023-38313-y. PMID 37147320